CLINICAL TRIAL: NCT03736200
Title: Neuro-rehabilitation Training Effects on Motion and Quality of Life After Acute Stroke and Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Principal Investigator, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKEB008/2018
Record Dates: First submitted 2018-11-01; First posted 2018-11-09 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2018-09

CONDITIONS: Stroke
Keywords: balance; movement; exergaming; posture; quality of life; gait
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exergaming 1/day (Active Comparator): Post stroke group that received 4 weeks of intensive therapy. (1/day)
  Interventions: Other: Exergaming group
- physiotherapy (Active Comparator): Post stroke group that received 4 weeks of traditional physiotherapy.
  Interventions: Other: Physiotherapy
- Exergaming 2/day (Active Comparator): Post stroke group that received 4 weeks of intensive therapy. (2/day)
  Interventions: Other: Exergaming group 2/day

INTERVENTIONS:
Other: Exergaming group — Neurorehabilitation - 4-week-long intervention, targeted postural instability and mobility using at-limit intensity sensori and visuomotor agility training. (1/day)
  Other Names: EXE group
  Arms: Exergaming 1/day
Other: Physiotherapy — Physiotherapy 4-week-long.
  Other Names: Physio group
  Arms: physiotherapy
Other: Exergaming group 2/day — Neurorehabilitation - 4-week-long intervention, targeted postural instability and mobility using at-limit intensity sensori and visuomotor agility training. (2/day)
  Other Names: EXE2 group
  Arms: Exergaming 2/day

SUMMARY:
High intensity motion improves motor functions and quality of life in a neurologist. The investigators want to improve the clinical condition and quality of life of post-STROKE participants with a special sensory motor and visual motor agility therapy.

DETAILED DESCRIPTION:
High intensity motion improves engine function and quality of life in a neurologist. With special sensory motor and visual motility, investigaters want to improve the clinical condition and quality of life of STROKE participants.

The investigaters randomly select participants who only perform the rehabilitation treatment have performed. The other group that will receive the study's control group will receive the traditional rehabilitation physiotherapy treatment.

The investigaters assess the condition and quality of life of the patients. (EQ5-D, Barthel index, MRS test) The ivestigaters examine the functional movement and equilibrium variables of patients. (6MWT, Berg balance test, postgraduation) After that, participants are undergoing a 4-week intensive rehabilitation treatment. All participants are in post stroke.

Primary Hypothesis will be changes in life-quality tests (EQ5-D, Barthel index, MRS test). Functional tests show progress 6MWT, Berg balance test and postural control testing with posturography. The results are compared and evaluated among the groups.

The expected hypothesis is that visual and acoustic stimulation produces a better physical state at higher intensity.

ELIGIBILITY:
Inclusion Criteria:

* post stroke
* 6MWT : 120>
* minimum after stroke 2 weeks

Exclusion Criteria:

* Sever heart problem
* sever demeanor
* alcoholism
* drug problems

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Quality of life measured by Barthel index | 4 weeks
  questionnaire
gait / functional test | 4 weeks
  6 minute walk test (m)
balance test | 4 weeks
  Berg balance test
postrural control test | 4 weeks
  posturography (mm)
Quality of life measured by EQ5-D scale | 4 weeks
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- József Tollá, Kaposvár, Somogy County, Hungary

REFERENCES:
- [Derived] Tollar J, Nagy F, Csutoras B, Prontvai N, Nagy Z, Torok K, Blenyesi E, Vajda Z, Farkas D, Toth BE, Repa I, Moizs M, Sipos D, Kedves A, Kovacs A, Hortobagyi T. High Frequency and Intensity Rehabilitation in 641 Subacute Ischemic Stroke Patients. Arch Phys Med Rehabil. 2021 Jan;102(1):9-18. doi: 10.1016/j.apmr.2020.07.012. Epub 2020 Aug 27. PMID 32861668
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=stroke+virtual+reality